CLINICAL TRIAL: NCT03737331
Title: Variable Visual Stimulus as a Novel Approach for Gait Rehabilitation
Acronym: VISNA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Canceled
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0395-18-FB
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Gait Disorders, Neurologic
Keywords: Visual; Variability; Gait; Fractals; Rehabilitation; Brain
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Older adults at risk of a fall will participate in an 8-week training program. There will be four groups: no stimulus (i.e., control), invariant, random and variable stimuli. The training program will consist in an 8-week program, 3 sessions per week. For each training session, participants will come to the Biomechanics Research Building for a 30-minute training session (2 x 10-minute walking trials with a 10-minute resting period in between), 3 times per week. During the training session, the subjects will be instructed to walk while viewing and synchronizing the steps with the visual stimulus. In the first session of weeks 3, 5 and 7, the subjects will undergo a reassessment of the preferred stride time, wearing the footswitches. This reassessment will be needed to recalculate the preferred stride time and incorporate it in the stimulus in use, in case it has been changed as an effect of the training.
Who Masked: Participant
Masking Description: Participants will be randomly assigned with a block randomization design for one of the four groups: no stimulus (i.e. control), invariant, random and variable stimuli. Subjects will be assigned to unique ID code such as 'S00NC', where S means subject, 00N refers to participant number (i.e., 001 or 100), and C the group condition (N - No stimulus; P - Periodic stimulus; V - Variant stimulus; R - Random stimulus).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fractal visual cueing (Experimental): This stimulus will consist of a visual moving bar displayed on a small monitor attached to a pair of glasses. The temporal structure of the movement will be fractal (i.e., pink noise). Participants will be asked to match their hell strikes of right foot with the top of the moving bar's path and their heel strikes of left foot to the bottom.
  Interventions: Behavioral: Fractal visual cueing
- Periodic visual cueing (Active Comparator): This stimulus will consist of a visual moving bar displayed on a small monitor attached to a pair of glasses. The temporal structure of the movement will be periodic (i.e., invariant). Participants will be asked to match their hell strikes of right foot with the top of the moving bar's path and their heel strikes of left foot to the bottom.
  Interventions: Behavioral: Periodic visual cueing
- Random visual cueing (Sham Comparator): This stimulus will consist of a visual moving bar displayed on a small monitor attached to a pair of glasses. The temporal structure of the movement will be random (i.e., white noise). Participants will be asked to match their hell strikes of right foot with the top of the moving bar's path and their heel strikes of left foot to the bottom.
  Interventions: Behavioral: Random visual cueing
- Control (No Intervention): Natural walking.

INTERVENTIONS:
Behavioral: Fractal visual cueing — Walking to an external visual fractal (i.e., pink noise) stimulus.
  Arms: Fractal visual cueing
Behavioral: Periodic visual cueing — Walking to an external visual periodic (i.e., invariant) stimulus.
  Arms: Periodic visual cueing
Behavioral: Random visual cueing — Walking to an external visual random (i.e., white noise) stimulus.
  Arms: Random visual cueing

SUMMARY:
Deterioration in walking performance as a result of disease or simply as a result of aging is a serious threat to independence in older adults. In this project, the investigators propose an innovative visual stimulus, based on advanced mathematical and biological theories, with which older adults can walk in time to improve their walking. The investigators' goal is to apply this simple, cost-effective, and novel gait rehabilitation therapy across all populations who have difficulties walking, e.g. stroke patients, fallers or those who undergo joint replacement.

DETAILED DESCRIPTION:
Walking synchronized to a visual stimulus is commonly used for gait rehabilitation, and has been shown to alter gait parameters such as stride length and stride time in a variety of patient populations. Typically, the patient is instructed to walk by stepping on lines or other markers placed on the ground presented in a fixed, invariant distance with each other. Whilst improvements in gait parameters have been observed in these experimental conditions, the investigators submit that a fundamentally different approach could lead to much greater benefits. The investigators' laboratory has successfully shown that walking to an invariant stimulus, with no variability, runs contrary to the natural stride-to-stride fluctuations (i.e., gait variability) that are known to exist in human gait. The investigators propose that the elimination of variability from gait, as is the case when walking with invariant external cueing, will not provide the movement abilities needed by individuals with reduced mobility to navigate the real world, unpredictable environments. In this project, the investigators propose an alternative approach to rehabilitation of gait disorders with respect to external cueing that takes the natural variability of healthy gait into account. The investigators have previously shown that young and older adults when walking to an invariant stimulus, display diminished natural stride-to-stride fluctuations. Preliminary data has also shown that the natural stride-to-stride fluctuations that exist in healthy gait are altered with aging, but can also be restored to levels similar to young adults when walking to a Variable Visual Stimulus. The investigators proposed solution is then to transform the standard invariant visual cueing paradigm by using a Variable Visual Stimulus that reflects the variable movement patterns found in healthy gait. This is because the presentation of our Stimulus will be variable, but it will not be random. There will be a pattern contained within the presentation of our Stimulus that is based upon the patterns found in healthy young adults. This project will investigate the long-term effects of viewing an invariant, a random and a variable visual stimulus on gait variability in older adults. Furthermore, the investigators will investigate the retention effects at 1- and 3-months of an 8-week program. The central hypothesis is that older adults who are at risk of falling will demonstrate greater improvements in gait variability and adaptive gait tasks when walking with a Variable Visual Stimulus that reflects the variable movement patterns found in healthy gait. The impact of this project will be transformational regarding gait rehabilitation for older adults who are at risk of falls. This simple, cost-effective method would be accessible to all gait rehabilitation clinics requiring only ubiquitously available glasses.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide informed consent.
* Be able to walk independently without an assistive device.
* Not suffer from neurological disease.
* Not suffer from any lower limb disabilities, injuries or disease.

Exclusion Criteria:

* If diagnosed with a pathology that directly affects the musculoskeletal system such as rheumatoid arthritis, neuropathy or myopathy, vertigo, joint replacement, diabetes, stroke or other vascular problems, scoliosis, uncorrected vision problems,major surgery in the last 6 months, or acute illness.
* Any neurologic conditions or lower limb disabilities or disease.
* History of seizures, migraines or headaches, or are visually impaired.
* Subjects unable to walk unassisted or unable to perform 10 minutes of continuous walking.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Stride length | Through study completion, an average of 1 year
  Meters
Stride time | Through study completion, an average of 1 year
  Seconds
Stride speed | Through study completion, an average of 1 year
  Meters/seconds
Cortical hemodynamics | Through study completion, an average of 1 year
  Micromoles

SECONDARY OUTCOMES:
Joint angles | Through study completion, an average of 1 year
  Radians
Peak torque of knee extensor muscles at 60º/s | Through study completion, an average of 1 year
  Newton-meters

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Silva, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stergiou N, Decker LM. Human movement variability, nonlinear dynamics, and pathology: is there a connection? Hum Mov Sci. 2011 Oct;30(5):869-88. doi: 10.1016/j.humov.2011.06.002. Epub 2011 Jul 29. PMID 21802756
- [Background] Brach JS, Wert D, VanSwearingen JM, Newman AB, Studenski SA. Use of stance time variability for predicting mobility disability in community-dwelling older persons: a prospective study. J Geriatr Phys Ther. 2012 Jul-Sep;35(3):112-7. doi: 10.1519/JPT.0b013e318243e5f9. PMID 22314273
- [Background] Brach JS, Studenski S, Perera S, VanSwearingen JM, Newman AB. Stance time and step width variability have unique contributing impairments in older persons. Gait Posture. 2008 Apr;27(3):431-9. doi: 10.1016/j.gaitpost.2007.05.016. Epub 2007 Jul 13. PMID 17632004
- [Background] Brach JS, Lowry K, Perera S, Hornyak V, Wert D, Studenski SA, VanSwearingen JM. Improving motor control in walking: a randomized clinical trial in older adults with subclinical walking difficulty. Arch Phys Med Rehabil. 2015 Mar;96(3):388-94. doi: 10.1016/j.apmr.2014.10.018. Epub 2014 Nov 10. PMID 25448244
- See also: Kaipust JP, McGrath D, Mukherjee M, Stergiou N. Gait variability is altered in older adults when listening to auditory stimuli with differing temporal structures. Ann Biomed Eng. 2013;41(8):1595-1603. doi:10.1007/s10439-012-0654-9. — https://link.springer.com/content/pdf/10.1007%2Fs10439-012-0654-9.pdf